CLINICAL TRIAL: NCT03204409
Title: Longitudinal Clinical and Virological Study Among Symptomatic Patients With Zika Virus Infection in the City of Sao Paulo, Brazil
Brief Title: ZIKAlliance Natural History Study
Acronym: ZIKAllianceNH
Status: Withdrawn | Type: Observational
Why Stopped: No ZIKA cases at study site
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thomas Jaenisch, Senior Scientist, University of Heidelberg Medical Center
Other Study IDs: 734548NH (EC | H2020 | RIA)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Zika Virus; Zika Virus Infection
Keywords: CHIKV; DENGUE; Chikungunya; DENV
MeSH Terms: conditions — Zika Virus Infection; Dengue; Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, urine and genital fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic adults: adult patients (>18 years) presenting with febrile or rash illness of short duration (<72h)

SUMMARY:
Study to enroll up to 1000 adult patients (>18 years) presenting with febrile or rash illness of short duration (<72h) in designated clinics in the State of Sao Paulo, Brazil.

DETAILED DESCRIPTION:
* Study to enroll up to 1000 adult patients (>18 years) presenting with febrile or rash illness of short duration (<72h) in designated clinics in the State of Sao Paulo, Brazil.
* Following enrolment (day 0), patients will be followed up at days 2-3, 7, 14, 21, 30, 90, 180 and 360 with clinical and biological procedures (blood and urine samples).
* For patients with proven ZIKA Virus (ZIKV) infection, follow-up samples will include blood, saliva, urine and genital samples.
* For non-ZIKV infected patients, follow-up samples will include serological monitoring at days 14, 30, 180 and 360, and for men, possible assessment of genital fluids at day 180.
* All patients will be evaluated for impact on disability up to one year. Household adult contacts of ZIKV patients will be invited for ZIKV evaluation including collection of blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Rash or Fever illness
* within 72 hours of symptom onset

Exclusion Criteria:

* presence of symptoms or complications indicative of a bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Population
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
ZIKA Virus Infection | up to one year
  Clinical Characterization
DENGUE Virus Infection | up to one year
  Clinical Characterization
Chikungunya Virus Infection | up to one year
  Clinical Characterization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jänisch, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avelino-Silva VI, Mayaud P, Tami A, Miranda MC, Rosenberger KD, Alexander N, Nacul L, Segurado A, Pohl M, Bethencourt S, Villar LA, Viana IFT, Rabello R, Soria C, Salgado SP, Gotuzzo E, Guzman MG, Martinez PA, Lopez-Gatell H, Hegewisch-Taylor J, Borja-Aburto VH, Gonzalez C, Netto EM, Saba Villarroel PM, Hoen B, Brasil P, Marques ETA, Rockx B, Koopmans M, de Lamballerie X, Jaenisch T; ZIKAlliance Clinical Study Group. Study protocol for the multicentre cohorts of Zika virus infection in pregnant women, infants, and acute clinical cases in Latin America and the Caribbean: the ZIKAlliance consortium. BMC Infect Dis. 2019 Dec 26;19(1):1081. doi: 10.1186/s12879-019-4685-9. PMID 31878895